CLINICAL TRIAL: NCT06988852
Title: Conversion Treatment With Hepatic Arterial Infusion of Oxaliplatin, Leucovorin and Fluorouracil Plus Intravenous Bevacizumab or Cetuximab for Initially Unresectable Colorectal Liver Metastasis: A Prospective Study
Brief Title: FOLFOX-HAIC as Conversion Treatment for Initially Unresectable Colorectal Liver Metastasis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Chen Xiaoping, Professor, Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHALLENGE-A1
Record Dates: First submitted 2025-05-04; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Liver Metastasis (CRLM)
MeSH Terms: interventions — Folfox protocol; Oxaliplatin; Leucovorin; Fluorouracil; Bevacizumab; Cetuximab; Hepatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Patients in the treatment group would undergo FOLFOX-HAIC combining Bevacizumab or Cetuximab
  Interventions: Combination Product: FOLFOX (oxaliplatin, leucovorin, 5-fluorouracil [5FU]); Procedure: hepatic arterial infusion chemotherapy (HAIC); Drug: Bevacizumab; Drug: Cetuximab (Erbitux); Procedure: liver resection

INTERVENTIONS:
Combination Product: FOLFOX (oxaliplatin, leucovorin, 5-fluorouracil [5FU]) — The procedures of FOLFOX-HAIC were as follows: 1) a 5 French sheath was inserted into the femoral artery by Seldinger technique, then a 3.5 French catheter entered the coeliac trunk and superior mesenteric artery to assess the feeding arteries of tumors and identify any extra-collateral vessels which may cause drug leakage. These vessels would be embolized with gelatin sponge particles or metallic coils if necessary. A 2.7 French microcatheter was selectively inserted into the left/right/proper hepatic artery then patients were transferred to inpatient ward to start chemotherapy drug infusion. The FOLFOX regimen involving oxaliplatin (130mg/m2, day 1, 0-2h), leucovorin (400 mg/m2, day 1, 2-3h), 5-Fu (400mg/m2, day 1, bolus at 3h, then 2400 mg/m2, day 1-3, 3-49h), was administered via the microcatheter. The microcatheter and sheath were removed after HAIC finished. We didn't implanted port catheter system and repeated percutaneous femoral artery puncture and catheterization once every 3
Procedure: hepatic arterial infusion chemotherapy (HAIC) — The procedures of FOLFOX-HAIC were as follows: 1) a 5 French sheath was inserted into the femoral artery by Seldinger technique, then a 3.5 French catheter entered the coeliac trunk and superior mesenteric artery to assess the feeding arteries of tumors and identify any extra-collateral vessels which may cause drug leakage. These vessels would be embolized with gelatin sponge particles or metallic coils if necessary. A 2.7 French microcatheter was selectively inserted into the left/right/proper hepatic artery then patients were transferred to inpatient ward to start chemotherapy drug infusion.
Drug: Bevacizumab — We would inject bevacizumab at the dose of 7.5mg/kg once every 3 weeks if the primary tumors located from right-side to splenic flexure colon or the genotype of RAS or RAF was mutational.
Drug: Cetuximab (Erbitux) — We would inject cetuximab at an initial dose of 400mg/m2 and maintained a dose of 250mg/m2 once every week if we didn't choose bevacizumab.
Procedure: liver resection — If patients reached potential resectable state, we would perform liver resection.

SUMMARY:
Try FOLFOX-HAIC combining bevacizumab or cetuximab for initially unresectable colorectal liver metastasis patients to increase the conversion to resection rate to improve long-term survival outcomes

DETAILED DESCRIPTION:
Colorectal cancer (CRC) was a common malignancy. Approximately 50% CRC patients would develop either synchronous or metachronous liver metastasis, which served as the leading cause of death in CRC, during the course of their diseases. Complete resection of all liver metastases is a major contributor to long-term survival with a median OS of 35 months, while it is just 20-24 months in modern chemotherapy. However,80%-90% colorectal liver metastasis (CRLM) patients present with initially unresectable diseases and the median OS in untreated patients is only 7.5 months. Liver transplantation achieves a 5-year OS rate of 56% compared to the rate of 9% for systemic chemotherapy, organ shortage and high cost limit its popularization. Conversion treatment refers to applying local and/or systemic treatment for IU-CRLM to eliminate technical or biologic unresectable factors to gain potential resectable states and is associated with a 5-year OS rate of 30%-61% in successful patients, which is non-inferior to those who are initially resectable. However, the conversion to resection rates (CTRRs) with negative margin vary from 1.7% to 66% depending on treatment regimens. So, promoting the conversion ability is the only way to improve long-term survival.

The systemic conversion treatment includes systemic chemotherapy and target agents. It shows high adverse event (AE) rates in practice and the CTRRs varies from 1.7% to 49%, which is unsatisfactory. The locoregional conversion treatment, such as hepatic arterial infusion chemotherapy (HAIC), transarterial chemoembolization (TACE), transarterial radioembolization (TARE) and so on, is only suitable for liver-only metastases. For the reason of CRLM deriving predominant blood supply from hepatic artery while liver parenchyma mainly from portal vein, transarterial interventional therapy may not only improve the CTRRs but also reduce AE rates. It's a pity that the CTRRs in TACE or TARE only range from 7% to 10%. HAIC achieves 17.8%-66% CTRRs depending on different drug regimens. Target agents indeed increases the CTTRs in systemic chemotherapy, but bevacizumab doesn't increases it in FUDR-HAIC and brings unexpectedly biliary toxicity. However, in unresectable hepatocellular carcinoma (uHCC), FOLFOX-HAIC combining with Sintilimab® and bevacizumab achieved a CTRR of 48.2% and no biliary toxicity event occurred. Another study, oxaliplatin-HAIC with systemic chemotherapy plus cetuximab achieved an impressive CTTR of 66% but was only suitable for patients without mutational RAS. Maybe a new regimen, oxaliplatin-based complete arterial infusion regimen combining with bevacizumab or cetuximab for IU-CRLM could achieve a milestone outcome, but no literature had reported it.

In this study, we establish a prospective and consecutive IU-CRLM patient cohort treated with FOLFOX-HAIC combining with bevacizumab or cetuximab to evaluate the CTRR, tumor response, safety and long-term oncological outcomes.

ELIGIBILITY:
Inclusion Criteria:

* age 18-75 years
* no history of other malignant diseases
* refuse or progress in prior systemic treatment
* diagnosed as CRLM confirmed by pathology, in spite of whether the primary tumor had been resected
* at least one lesion in the liver could be measured
* left ventricular ejection ≥45%, forced expiratory volume in one second/forced vital capacity≥60% and Eastern Cooperative Oncology Group (ECOG) score of 0-1
* Child-Pugh class A
* adequate organ function, i.e.: white blood cell (WBC) ≥3.0×109/L, neutrophils ≥1.5×109/L, platelet (PLT) ≥75×109/L, total bilirubin ≤30μmol/L, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤200U/L, creatinine ≤150μmol/L

Exclusion Criteria:

* extra-hepatic metastasis verified by medical imaging
* unable to tolerate chemotherapy, anesthesia or surgery
* allergy or previous intolerable to any agent of oxaliplatin, leucovorin, 5-Fu, bevacizumab or cetuximab
* tumor spread in abdomen
* cerebral infarction, cerebral hemorrhage, gastrointestinal hemorrhage/perforation within 6 months, coagulation disorders and gastrointestinal ulcer
* primary tumor may not be completely resected
* prior treatment of CRLM with resection, ablation or radiation
* incomplete clinical or follow-up data

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
conversion to resection rate | 180 days
  conversion to resection rate: the number of patients underwent liver resection/total patients underwent FOLFOX-HAIC combining with target agents

SECONDARY OUTCOMES:
drug treatment safety assessment | Baseline up to study termination, assessed up to 12 months.
  Any adverse event during treatment that is incompatible with the therapeutic purpose of the medication. The incidence and severity of adverse events and serious adverse events as assessed according to CTCAE v5.0.
objective response rate | From the time of enrollment until disease progression, death, or the end of the study, assessed up to 12 months.
  Objective response rate (ORR) was defined as the sum of cases with complete response (CR) and partial response (PR) which assessed by the RECIST 1.1 criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No